CLINICAL TRIAL: NCT06431178
Title: A Comparative Study Between General Anesthesia Versus Sedation By Dexmedetomidine and Ketamine With Local Infiltration for Percutaneous Transcatheter Closure of Atrial Septal Defect in Pediatric Patients
Brief Title: General Anesthesia Versus Sedation By Dexmedetomidine and Ketamine With Local Infiltration for Percutaneous Transcatheter Closure of Atrial Septal Defect in Pediatric Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Aya Ebrahim Abdelhafez Mashal, Assistant Lecturer of Anesthesiology, Surgical Intensive Care and Pain Medicine, Faculty of Medicine, Tanta University, Tanta, Egypt., Tanta University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 36264MD57/3/23
Record Dates: First submitted 2024-05-13; First posted 2024-05-28 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: General Anesthesia; Dexmedetomidine; Ketamine; Local Infiltration; Atrial Septal Defect
MeSH Terms: conditions — Heart Septal Defects, Atrial | interventions — Anesthesia, General; Anesthesia, Local

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- General anesthesia (Active Comparator): General anesthesia will be induced by 6% sevoflurane with a face mask. An intravenous line(22-g cannula )will be inserted then fentanyl 1mcg-kg will be given . Endotracheal tube will be used to intubate the patient .Anesthesia will be maintained by 2%sevoflurane inhalation in an oxygen air compination 1:1 throught the operation.
  Crystalloid solution was used to replenish fluid according "4/2/1-rule". Monitoring during the procedure include , ejection fraction (EF),blood pressure, heart rate, respiratory rate, and O2 saturation are measured at baseline, after induction, 10 min after catheter insertion,30 min during procedure and post emergence.
  Interventions: Other: General Anesthesia
- Local anesthesia (Experimental): A nasal cannula was placed and oxygen delivered at 2 to 3 L/minute. An intravenous line will be inserted (22-g cannula). The sedation regimen will include loading dose of dexmedetomidine (1 mcg/kg) and ketamine (1mg/kg) over 10 minutes . The patient will receive an infusion of dexmedetomidine at 0.7 mcg/kg per hour and ketamine 0.5 mg/kg/hr as maintenance sedation .Local infilteration of xylocaine 2% at dose 2mg/kg will be given for vascular access in cardiac catheterization . After completion of the procedure the infusion pump will be stopped to ensure that the patient is fully awake and vitally stable
  Interventions: Other: Local anesthesia

INTERVENTIONS:
Other: General Anesthesia — General anesthesia will be induced by 6% sevoflurane with a face mask. An intravenous line(22-g cannula )will be inserted then fentanyl 1mcg-kg will be given . Endotracheal tube will be used to intubate the patient .Anesthesia will be maintained by 2%sevoflurane inhalation in an oxygen air compination 1:1 throught the operation . Crystalloid solution was used to replenish fluid according "4/2/1-rule". Monitoring during the procedure include , ejection fraction (EF),blood pressure, heart rate, respiratory rate, and O2 saturation are measured at baseline, after induction, 10 min after catheter insertion,30 min during procedure and post emergence.
  Arms: General anesthesia
Other: Local anesthesia — A nasal cannula was placed and oxygen delivered at 2 to 3 L/minute. An intravenous line will be inserted (22-g cannula). The sedation regimen will include loading dose of dexmedetomidine (1 mcg/kg) and ketamine (1mg/kg) over 10 minutes . The patient will receive an infusion of dexmedetomidine at 0.7 mcg/kg per hour and ketamine 0.5 mg/kg/hr as maintenance sedation .Local infilteration of xylocaine 2% at dose 2mg/kg will be given for vascular access in cardiac catheterization . After completion of the procedure the infusion pump will be stopped to ensure that the patient is fully awake and vitally stable
  Arms: Local anesthesia

SUMMARY:
The aim of the present study is to compare between general anesthesia versus sedation with dexmedetomidine and ketamine with local infilteration at the catheter insertion site in pediatric patients undergoing transcutaneous closure of atrial septal defect on hemodynamic changes.

DETAILED DESCRIPTION:
Atrial septal defect (ASD) is one of the most common types of congenital heart defects, occurring in about 25% of children General anaesthesia is usually obtained with tracheal intubation and mechanical ventilation or spontaneous breathing, the depth of anesthesia required to tolerate the presence of a tracheal tube will invariably lead to some reduction in myocardial contractility and alteration of respiratory mechanics. The goal of anesthetic technique is to provide sedation and analgesia during cardiac catheterization to ensure immobility and hemodynamic stability.

Ketamine is an N-methyl-D-aspartate receptor (NMDA) antagonist with sedative, analgesic, and sympathomimetic effects. Among its benefits ,it has the ability to protect airway reflexes with minimal effect on ventilatory drive.

Dexmedetomidine is a highly selective alpha-2 adrenoreceptor agonist with sedative, anxiolytic, and analgesic effect, it also blunts the sympathetic nervous system response to surgical stimulation.

ELIGIBILITY:
Inclusion Criteria:

* Aged 3-8 years old.
* Both genders.
* American Society of Anesthesiologists (ASA) physical status II-III
* Pediatric patients scheduled for elective transcatheter atrial septal defect closure.

Exclusion Criteria:

* Patients with multiple congenital anomalies.
* Patients with congestive heart failure
* Patients with Organ dysfunction liver or renal disease or pulmonary disease.
* Recent chest infection.
* Airway abnormalities.

Ages: 3 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
Heart rate | Immediately after the intervention
  Heart rate will be measured at baseline, after induction ,10 min after catheter insertion site,30 min during procedure and post emergence in both groups.

SECONDARY OUTCOMES:
Mean arterial blood pressure | Immediately after the intervention
  Mean arterial blood pressure will be measured at baseline, after induction ,10 min after catheter insertion site,30 min during procedure and post emergence in both groups.
O2 saturation | Immediately after the intervention
  O2 saturation will be measured at baseline, after induction ,10 min after catheter insertion site,30 min during procedure and post emergence in both groups.
Respiratory rate | Immediately after the intervention
  Respiratory rate will be measured at baseline, after induction ,10 min after catheter insertion site,30 min during procedure and post emergence in both groups.
Lengh of hospital stay | 28 days postoperative
  Length of hospital stay will be measured from admission till discharge from hospital
Recovery time | Immediately after discharge from post-anesthesia care unit
  Recovery time will be measured from the end of surgery till discharge from post-anesthesia care unit (PACU).
Complications | 24 hours postoperative
  Postoperative complications such as arrythmia, hypotension, bradycardia, nausea and vomiting will be measured.

CONTACTS AND LOCATIONS:
Locations (1):
- Aya Ebrahim Abdelhafez Mashal, Tanta, El-Gharbia Governorate, Egypt, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author